CLINICAL TRIAL: NCT04494490
Title: Resolving the Burden of Low Back Pain in Military Service Members and Veterans: A Pragmatic Clinical Trial
Acronym: RESOLVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Gorczynski (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); University of Pittsburgh (Other); Naval Health Research Center (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); VA New York Harbor Healthcare System (U.S. Federal Agency); Marine Corps Base Camp Pendleton (Other)
Responsible Party: Sponsor-Investigator, Sara Gorczynski, Site Principal Investigator, United States Naval Medical Center, San Diego
Organization: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NMCSD.2018.0034
Record Dates: First submitted 2020-07-13; First posted 2020-07-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Condition (No Intervention): During the usual care condition the therapists will be instructed "to act as usual," that is, to read the guidelines on low back pain if they have read previous published guidelines and not read these guidelines if they have not read any other guidelines.
- CPG+PIPT Condition (Active Comparator): An active Clinical Practice Guidelines (CPG) implementation strategy will be utilized with an education component in Psychologically Informed Physical Therapy (PIPT) with peer opinion leaders and a monthly audit/feedback on CPG adherence rates and patient outcomes
  Interventions: Behavioral: Clinical Practice Guidelines and Psychologically Informed Physical Therapy training/audit/feedback

INTERVENTIONS:
Behavioral: Clinical Practice Guidelines and Psychologically Informed Physical Therapy training/audit/feedback — The aim of the active training strategy is to improve the knowledge and skills of physical therapists with regard to evidence-based physical therapy with an emphasis on active treatments and PIPT for the treatment of patients with low back pain and to encourage increased adherence with CPGs. This Continuing Education (CE) training session will be offered to all therapists regardless of study participation. During the CE training session, focus will be placed on interventions that have been shown to be effective, such as interactive education and discussion, feedback, and reminders.
  Arms: CPG+PIPT Condition

SUMMARY:
The RESOLVE trial will provide a pragmatic approach to evaluate whether Physical Therapy Clinical Practice Guideline adherence can reduce pain, disability and downstream healthcare utilization for low back pain within the Departments of Defense and Veterans Affairs healthcare systems.

DETAILED DESCRIPTION:
Physical therapy (PT) is frequently used for the management of low back pain (LBP) within the U.S. Departments of Defense (DoD) and Veterans Affairs (VA). However, variations in PT practice patterns and utilization of ineffective interventions lower the quality and increase the cost of care. Although, adherence to the clinical practice guidelines (CPGs) can improve outcomes and cost effectiveness of LBP care, PT CPG adherence rates remain below 50%. The RESOLVE trial will evaluate the effectiveness of an active PT CPG implementation strategy using an education/audit/feedback model for reducing pain, disability, medication use and cost of LBP care within the DoD and VA healthcare systems. The RESOLVE trial will include 3300 to 7260 patients with LBP from five DoD and VA medical facilities, using a stepped-wedge study design. An education/audit/feedback model will be used to encourage the physical therapists to better adhere to the PT CPG recommendations. The primary outcomes of disability and pain intensity will be measured with the Oswestry Disability Index and the Defense and Veterans Pain Rating Scale. Secondary outcomes will include the LBP-related medical resource utilization and biopsychosocial predictors of PT outcomes. Statistical analyses will be based on intention to treat principles and will use linear mixed models to compare treatment conditions, and examine the interactions between treatment and sub-grouping status. The RESOLVE trial will provide a pragmatic approach to evaluate whether PT CPG adherence can reduce pain, disability and downstream healthcare utilization for LBP within the DoD and VA healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Receiving physical therapy care for low back pain in an outpatient physical therapy setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4039 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Every two weeks over course of PT treatment, up to 12 weeks
  Change in Defense and Veterans Pain Rating Scale (DVPRS) score
Disability | Every two weeks over course of PT treatment, up to 12 weeks
  Change in Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Healthcare Utilization | One year
  Change in frequency of healthcare utilization:The medical resources of interest for this trial will include: 1) referrals to specialists (e.g., orthopedists, spine surgeons, physiatrists) and other health care providers, and 2) tests (e.g., x-rays, MRIs), surgical procedures (e.g., epidural steroid injections, laminectomy).
Healthcare Utilization | One year
  Change in extent of healthcare utilization:The medical resources of interest for this trial will include: 1) referrals to specialists (e.g., orthopedists, spine surgeons, physiatrists) and other health care providers, and 2) tests (e.g., x-rays, MRIs), surgical procedures (e.g., epidural steroid injections, laminectomy).
Analgesic Medication Use | One year
  Change in frequency of analgesic medication use: prescribing patterns for key drug classes commonly used for low back pain management such as non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen (Tylenol), opioid analgesics, skeletal muscle relaxants, antidepressants (e.g., tricyclic antidepressants and duloxetine), and drugs for neuropathic pain (e.g., gabapentin).
Analgesic Medication Use | One year
  Change in extent of analgesic medication use: prescribing patterns for key drug classes commonly used for low back pain management such as non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen (Tylenol), opioid analgesics, skeletal muscle relaxants, antidepressants (e.g., tricyclic antidepressants and duloxetine), and drugs for neuropathic pain (e.g., gabapentin).

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No